CLINICAL TRIAL: NCT05776446
Title: Retrospective Study on the Clinical Behavior of the Asqelio™ Trifocal Diffractive Intraocular Lens With Follow-up at 3 Months
Brief Title: Clinical Behavior of the Asqelio™ Trifocal Diffractive Intraocular Lens
Status: Completed | Type: Observational
Sponsor: AST Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASQT022022
Record Dates: First submitted 2023-02-13; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study was to evaluate distance, intermediate, and near vision in patients who have undergone cataract extraction with bilateral implantation of a new hydrophobic trifocal diffractive intraocular lens (IOL) with a biospheric design, the Asqelio Trifocal IOL (AST Products, Inc., Billerica MA, USA), along with patient-reported outcomes (PRO). For that purpose the clinical information of 50 eyes from 25 patients was retrospectively analyzed 3 months after implantation

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older submitted to cataract surgery with binocular implantation of Asqelio Trifocal TFLIO130C IOL
* Seeking spectacle independence after surgery
* IOL power between +5.0D y +34.0D
* Transparent ocular media, except for the cataract prior to surgery.
* Potential postoperatory visual acuity of 20/25 or better, as assessed prior to surgery

Exclusion Criteria:

* Preoperatory corneal astigmatism greater than 1.0D
* Previous corneal surgery or trauma
* Irregular cornea (e.g. keratoconus)
* Choroidal hemorrhage
* Microftalmos
* Severe corneal dystrophy
* Uncontrolled or medically controlled glaucoma
* Clinically significant macular changes
* Severe concomitant ocular condition
* Cataract not age-related
* Severe optic nerve atrophy
* Diabetic retinopathy
* Ambyopia
* Extremely shallow anterior chamber
* Severe chronic uveitis
* Pregnancy or lactating
* Rubella
* Mature/dense cataract difficulting preoperatory eye fundus assessment
* Previous retinal detachment
* Concurrent participation in another investigation involving drugs or medical devices

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are regular clinic patients submitted to bilateral conventional cataract surgery by phacoemulsification, who wanted to correct their refractive error and presbyopia, and thus were implanted with the trifocal IOL subject to study by common clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Uncorrected distance visual acuity | 3 months after implantation
  Uncorrected visual acuity for distance (4m) determined under photopic conditions using EDTRS optotypes, in LogMAR units
Best-corrected distance visual acuity | 3 months after implantation
  Best-corrected visual acuity for distance (4m) determined under photopic conditions using EDTRS optotypes, in LogMAR units
Uncorrected intermediate visual acuity | 3 months after implantation
  Uncorrected visual acuity for intermediate disntace (60cm) determined under photopic conditions using EDTRS optotypes, in LogMAR units
Distance-corrected intermediate visual acuity | 3 months after implantation
  Distance-corrected visual acuity for intermediate disntace (60cm) determined under photopic conditions using EDTRS optotypes, in LogMAR units
Uncorrected near visual acuity | 3 months after implantation
  Uncorrected visual acuity for near (40cm) determined under photopic conditions using EDTRS optotypes, in LogMAR units
Distance-corrected near visual acuity | 3 months after implantation
  Distance-corrected visual acuity for near (40cm) determined under photopic conditions using EDTRS optotypes, in LogMAR units
Defocus curve | 3 months after implantation
  Binocular defocus curve with best correction for distance obtained varying mergence from -4.0D to +2.0D in 0.5D steps

SECONDARY OUTCOMES:
Manifest Refraction | Preoperatively and 3 months after implantation
  Refraction determined monocularly by subjective refraction methods, in diopters
Adverse events | 3 months after implantation
  Percentage of subjects with adverse events (ocular and non ocular, severe and non severe), including secondary surgical interventions
Patient-reported outcomes CATQuest9SF | 3 months after implantation
  Patient reported outcomes were assessed by CATQuest9SF questionnaire
Patient-reported outcomes PRSIQ | 3 months after implantation
  Patient reported outcomes were assessed by patient-reported spectacle independence questionnaire (PRSIQ)
Patient-reported outcomes PRVSQ | 3 months after implantation
  Patient reported outcomes were assessed by the patient-reported visual symptoms questionnaire (PRVSQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital La Arruzafa, Córdoba, Cordoba, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cano-Ortiz A, Sanchez-Ventosa A, Gonzalez-Cruces T, Cerdan-Palacios D, Diaz-Mesa V, Gallego-Ordonez R, Galvez-Gomez T, Garcia Parrizas JA, Zurera Baena J, Villarrubia-Cuadrado A. Visual Performance, Satisfaction, and Spectacle Independence after Implantation of a New Hydrophobic Trifocal Intraocular Lens. J Clin Med. 2022 Oct 8;11(19):5931. doi: 10.3390/jcm11195931. PMID 36233798